CLINICAL TRIAL: NCT03752372
Title: Longitudinal Development of Intestinal Microbiome in IL10RA-deficient Patients After Hematopoietic Stem Cell Transplantation
Brief Title: Microbiome Alterations in IL10RA-deficient Patients After HSCT
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, The director of gastroenterology of Children's Hospital of Fudan University, Children's Hospital of Fudan University
Other Study IDs: HSCT microbiomte
Record Dates: First submitted 2018-11-19; First posted 2018-11-26 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Inflammatory Bowel Diseases; Microbiota
Keywords: interleukin 10 receptor alpha gene
MeSH Terms: conditions — Inflammatory Bowel Diseases; Inflammatory Bowel Disease 28, Autosomal Recessive | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HSCT cohort: IL10RA-deficient patients who received hematopoietic stem cell transplantation
  Interventions: Procedure: hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: hematopoietic stem cell transplantation — 1. Reduced intensity conditioning(RIC) chemotherapy regimen before transplantation
  2. All patients were cared for in single rooms ventilated with a highly effective particulate air filtration system. All patients received intravenous immunoglobulin and antimicrobial prophylaxis, which included antiviral, antifungal, and Pneumocystis jirovecii prophylaxis with ganciclovir and micafungin, as per routine clinical practice before transplantation.
  3. Umbilical cord blood transplantation

SUMMARY:
To elucidate the longitudinal development of intestinal microbiota in patients with IL10RA deficiency after hematopoietic stem cell transplantation (HSCT). The investigators planned to collect fecal samples from IL10RA-deficient patients who received HSCT. Samples were collected more than once every three days after engraftment in lamina flow ward and at least once a week before discharge. Microbial DNA was extracted from the fecal samples. And all analysis was based on the next generation sequencing data.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation is considered the only curative therapy for patients with interleukin-10 receptor-A(IL10RA) deficiency. The investigators aimed to collect the fecal samples of these patients throughout the conditioning, transplantation until discharge, providing a dense insight into the longitudinal development of intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* IL10RA gene mutations;
* Eligible for hematopoietic stem cell transplantation.

Exclusion Criteria:

* Unwilling to participate.

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients who were diagnosed with IL10RA deficiency and who received the hematopoietic stem cell transplantation in a tertiary hospital were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Shannon indices | during the hospitalization of each eligible patient, an average of 90 days per patient
  Shannon index is a popular diversity index in the ecological literature; minimum score is zero, higher values represent a better outcome
Simpson indices | during the hospitalization of each eligible patient, an average of 90 days per patient
  Simpson index in ecology is to measure the degree of concentration when individuals are classified into types; scale ranges [0,1]; lower values represent a better outcome
relative abundance of Proteobacteria | during the hospitalization of each eligible patient, an average of 90 days per patient
  describe the microbiome at the phylum level
relative abundance of Firmicutes | during the hospitalization of each eligible patient, an average of 90 days per patient
  describe the microbiome at the phylum level
Clostridium sensus_stricto_1 | during the hospitalization of each eligible patient, an average of 90 days per patient
  describe the microbiome at the genus level
Escherichia - Shigella | during the hospitalization of each eligible patient, an average of 90 days per patient
  describe the microbiome at the genus level

SECONDARY OUTCOMES:
chimerism | during the hospitalization of each eligible patient, an average of 90 days per patient
  The level of chimerism of each patient will be reported as percentages [0,100%]
manifestation of graft-versus-host disease | during the hospitalization of each eligible patient, an average of 90 days per patient
  describe the graft-versus-host disease happened to each patient
Sobs indices | during the hospitalization of each eligible patient, an average of 90 days per patient
  describe the the observed richness of each sample
Chao1 estimator | during the hospitalization of each eligible patient, an average of 90 days per patient
  describe the operational taxonomic unit(OTU) numbers of each sample
neutrophil cell count | during the hospitalization of each eligible patient, an average of 90 days per patient
  blood test results
platelet count | during the hospitalization of each eligible patient, an average of 90 days per patient
  blood test results

OTHER OUTCOMES:
relative abundance of Clostridiales | during the hospitalization of each eligible patient, an average of 90 days per patient
  describe the microbiome at the order level
Shannoneven indices | during the hospitalization of each eligible patient, an average of 90 days per patient
  measure the community evenness, scale ranges [0,1]; higher values represent a better outcome
Simpsoneven indices | during the hospitalization of each eligible patient, an average of 90 days per patient
  measure community evenness, scale ranges [0,1]; higher values represent a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, MD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peng K, Qian X, Huang Z, Lu J, Wang Y, Zhou Y, Wang H, Wu B, Wang Y, Chen L, Zhai X, Huang Y. Umbilical Cord Blood Transplantation Corrects Very Early-Onset Inflammatory Bowel Disease in Chinese Patients With IL10RA-Associated Immune Deficiency. Inflamm Bowel Dis. 2018 Jun 8;24(7):1416-1427. doi: 10.1093/ibd/izy028. PMID 29788474